CLINICAL TRIAL: NCT06293001
Title: Cross-Cultural Adaptation, Validity and Reliability of the Turkish Version of the Avoidance of Daily Activities Photo Scale for Patients With Shoulder Pain (ADAP Shoulder Scale)
Brief Title: Cross-Cultural Adaptation, Validity and Reliability of the Turkish Version of the ADAP Shoulder Scale
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, Associate Professor Elif TURGUT, Hacettepe University
Other Study IDs: SBA 23/349
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Questionnaire; Shoulder Pain; Validity; Reliability
Keywords: Questionnaire; Shoulder pain; Validity; Reliability; Cross-cultural adaptation
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with shoulder pain: Patients with shoulder pain, pain for at least three months and aged between 18 and 64 years, and for the re-test only participants with unchanged health status were included in the study. Patients with rheumatological, neurological or musculoskeletal diseases, invasive intervention in the last 3 months, active infection, history of cancer, post-traumatic condition requiring surgery were excluded.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Shoulder pain is a common musculoskeletal problem that increases disability and decreases quality of life in addition to socio-economic impact. Chronic pain is defined as pain lasting longer than three months. Chronic pain is a multidimensional and complex experience. According to this model, chronic pain is a multidimensional and complex experience. This experience may be accompanied by different pain beliefs, pain avoidance behaviours, pain-related fear of movement, anxiety and depression. Many conditions involving the shoulder complex including traumatic and non-traumatic pain, subacromial impingement, postoperative pain, rotator sheath tears, rotator sheath tendinopathy, shoulder arthritis, adhesive capsulitis, shoulder instabilities may lead to pain-related fear of movement.

Until now, pain-related fear and avoidance behaviours in patients with shoulder pain have been evaluated with the Tampa Kinesiophobia Scale, Pain Avoidance Beliefs Scale and Fear of Pain Scale. However, only patients with low back pain were included in the development of these scales. There was no scale developed specifically for shoulder pain. To fill this gap in the literature, Ansanello et al. developed the "Avoidance Daily Activities Photo Scale for Patients With Shoulder Pain (ADAP)" scale to evaluate pain avoidance behaviours in individuals with shoulder pain. Cross-cultural adaptation, validity and reliability of the Turkish version of the ADAP scale has not been studied.

The aim of our study was to perform cross-cultural adaptation, validity and reliability of the Turkish version of the Avoidance of Daily Activities Photo Scale for Patients with Shoulder Pain (ADAP Shoulder Scale).

DETAILED DESCRIPTION:
The research will be conducted at Hacettepe University Faculty of Physical Therapy and Rehabilitation, Athlete Health Unit. The research will be conducted according to the Consensus-Based Standards for the Selection of Health Measurement Instruments (COSMIN) guidelines.

Translation and cross-cultural adaptation of the ADAP Shoulder Scale will be carried out in five stages according to standard guidelines for scale translation and cross-cultural adaptation.It was planned to include 150 individuals with shoulder pain between the ages of 18 to 64 in the study.

The data collection for this planned study will be solely through surveys. The design of the study is a cross-sectional study aimed at developing and assessing the validity and reliability." Surveys specific to the research will be implemented in the study.

ELIGIBILITY:
Inclusion Criteria:

Patients with shoulder pain who have had pain for at least three months The ages between of 18 and 64.

Exclusion Criteria:

Rheumatological, neurological or musculoskeletal diseases, Non-invasive interventions performed in the last 3 months, Active infections, History of cancer, Conditions requiring post-traumatic surgery.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with shoulder pain were included in the study. Patients with shoulder pain, pain for at least three months and aged between 18 and 64 years, and for the re-test only participants with unchanged health status were included in the study. Patients with rheumatological, neurological or musculoskeletal diseases, invasive intervention in the last 3 months, active infection, history of cancer, post-traumatic condition requiring surgery were excluded.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Investigating Cross-Cultural Adaptation, Validity and Reliability of the Turkish Version of the Avoidance of Daily Activities Photo Scale for Patients with Shoulder Pain (ADAP Shoulder Scale) | 10 minutes
  A score of 0 represents the best score and a score of 10 represents the worst score and indicates worsening of the symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Turgut, Ass. Prof., Study Director — Hacettepe University
Locations (1):
- Elif Turgut, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No